CLINICAL TRIAL: NCT05524298
Title: Quality Of Life On Elderly Patients With Low Grade Non-Hodgkin Lymphoma Treated With Immunotherapy Or Immunochemotherapy And/Or Radiotherapy: An Observational Prospective Study Of The Fondazione Italiana Linfomi
Brief Title: Quality Of Life On Elderly Patients With Low Grade Non-Hodgkin Lymphoma
Status: Recruiting | Type: Observational
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Other Study IDs: FIL_QoL-ELDIND
Record Dates: First submitted 2022-07-29; First posted 2022-09-01 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Low Grade Non-Hodgkin's Lymphoma, Adult

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly Patients With Low Grade Non-Hodgkin Lymphoma: Elderly Patients With Low Grade Non-Hodgkin Lymphoma Treated With Immunotherapy Or Immunochemotherapy And/Or Radiotherapy.
  Assess QoL (quality of life) at baseline, at the end of treatment and after 1 year from the start of the therapy.

SUMMARY:
Aims of this study are to describe the variation of QoL (Quality of Life) during the clinical management of low-grade lymphoma in elderly subjects and to identify the most important factors at diagnosis and during treatment with an impact on QoL (Quality of Life).

DETAILED DESCRIPTION:
This is a prospective, multicenter, non-interventional study aiming at investigating on the changes in QoL (Quality of Life) during the clinical management of low-grade lymphoma in elderly subjects and to possibly identify the most important factors at diagnosis and during treatment with an impact on QoL (Quality of Life).

The study plans to enroll 150 patients with a local histologically confirmed diagnosis of indolent non-Hodgkin lymphoma fulfilling all the inclusion/exclusion criteria who provide written informed consent will be included in the study. Any type of treatment is allowed by the study (immunotherapy, immunochemotherapy at full or reduced dose, radiotherapy).

All patients must undergo Comprehensive Geriatric Assessment (CGA) before starting any protocol treatment.

Baseline, post-treatment and follow-up instrumental assessments and response evaluation is done as part of the routine clinical management for patients with indolent NHL (Non Hodgkin Lymphoma) . Response evaluation and all other assessments planned for the EOT (end of treatment) should be planned also in case of early withdrawal, according to clinical practice.

HRQoL (Health-related Quality of Life) evaluation will be done at time of informed consent form signature prior to treatment start, at the end of the treatment (ranging from 1 month to 6 months according to the duration of the treatment) and after 1 year from the start of the therapy.

QoL (quality of life) assessment includes all scales of the EORTC-QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of life Questionnaire-Core 30) and the FACT-Lym-LymS (Functional Assessment of Cancer Therapy - Lymphoma - lymphoma-specific symptoms questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* Local histological diagnosis of indolent B cell non-Hodgkin lymphoma: follicular lymphoma, marginal zone lymphoma (nodal, MALT (Mucosa-Associated Lymphoid Tissue), splenic), lymphoplasmacytic lymphoma/ Waldenström macroglobulinemia)
* Age ≥ 70 years
* Patient candidates to receive treatment for lymphoma
* Patient previously untreated for lymphoma
* Evaluation of Comprehensive Geriatric Assessment at baseline
* Ability to provide informed consent: subject understands and voluntarily signs an informed consent form approved by an IEC (Independent Ethics Committee), prior to registration into the study

Note: Patient treated in the context of a clinical trial is admitted

Exclusion Criteria:

* none

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly Patients With Low Grade Non-Hodgkin Lymphoma Treated With Immunotherapy Or Immunochemotherapy And/Or Radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
QoL (quality of life) scores at baseline - EORTC-QLQ-C30 | The endpoint wil be evaluated at the baseline.
  Quality of life is measured with the EORTC-QLQ-C30 (European Organisation for Research and Treatment of Cancer-Quality of life Questionnaire-Core 30) questionnaire)
QoL (quality of life) scores variations at the end of treatment - EORTC-QLQ-C30 | The endpoint will be evaluated from the beginning of the study to the end of therapy (up to 18 months)
  Quality of life is measured with the EORTC-QLQ-C30 (European Organisation for Research and Treatment of Cancer-Quality of life Questionnaire-Core 30)
QoL (quality of life) scores variations after 1 year from the start of therapy - EORTC-QLQ-C30 | The endpoint will be evaluated after 1 year from the start of therapy (up to 30 months)
  Quality of life is measured with the EORTC-QLQ-C30 (European Organisation for Research and Treatment of Cancer-Quality of life Questionnaire-Core 30) and FACT-Lym-LymS (Functional Assessment of Cancer Therapy - Lymphoma- lymphoma-specific symptoms questionnaire)
QoL (quality of life) scores at baseline - FACT-Lym-LymS | The endpoint wil be evaluated at the baseline.
  Quality of life is measured with the FACT-Lym-LymS (Functional Assessment of Cancer Therapy - Lymphoma- lymphoma-specific symptoms)
QoL (quality of life) scores variations at the end of treatment - FACT-Lym-LymS | The endpoint will be evaluated from the beginning of the study to the end of therapy (up to 18 months)
  Quality of life is measured with the FACT-Lym-LymS (Functional Assessment of Cancer Therapy - Lymphoma- lymphoma-specific symptoms questionnaire)
QoL (quality of life) scores variations after 1 year from the start of therapy - FACT-Lym-LymS | The endpoint will be evaluated after 1 year from the start of therapy (up to 30 months)
  Quality of life is measured with FACT-Lym-LymS (Functional Assessment of Cancer Therapy - Lymphoma- lymphoma-specific symptoms questionnaire)

SECONDARY OUTCOMES:
Overall Survival (OS) | The endpoint will be evaluated from the beginning to the end of the study (up to 30 months)
  Overall survival, the percentage of patients alive, is defined as the time between the date of registration and the date of death from any cause.
Progression-Free Survival (PFS) | The endpoint will be evaluated from the beginning to the end of the study (up to 30 months)
  Progression-Free Survival is defined as the time between the date of registration and the date of disease progression, relapse or death from any cause.
Event-Free Survival (EFS) | The endpoint will be evaluated from the beginning to the end of the study (up to 30 months)
  Event-Free Survival is defined as the time from start of treatment to disease progression, death or discontinuation of treatment for any reason (e.g. toxicity, patient preference), or initiation of a new treatment without document progression.
Overall Response Rate (ORR) | The endpoint will be evaluated from the beginning to the end of the study (up to 30 months)
  Overall response rate is defined as the proportion of patients who have a complete response (CR), or partial response (PR) or stable disease (SD) to therapy.Overall Response Rate (ORR) will be defined according to the Lugano 2014 criteria.
Registration of safety | The endpoint will be evaluated from the beginning to the end of the study (up to 30 months)
  Safety is defined as incidence, nature, and severity of adverse events graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), current version.

CONTACTS AND LOCATIONS:
Overall Officials: Salvatrice Mancuso, Principal Investigator — Ematologia - A.O.U. Policlinico Giaccone, Palermo
Locations (20):
- Italy (20):
  - S.C. Ematologia - A.O. SS. Antonio e Biagio e Cesare Arrigo, Alessandria, Alessandria
  - Clinica di Ematologia - A.O.U. Ospedali Riuniti, Ancona, Italy
  - U.O.C. Ematologia - IRCCS Istituto Tumori Giovanni Paolo II, Bari, Italy
  - Ematologia - ASST Spedali Civili di Brescia, Brescia, Italy
  - Ematologia - Ospedale di Castelfranco Veneto, Castelfranco Veneto, Italy
  - U.O.C. di Ematologia - Azienda Ospedaliera Universitaria Policlinico - Rodolico S. Marco, Catania, Italy
  - Unità funzionale di Ematologia - Azienda Ospedaliera Universitaria Careggi, Florence, Italy
  - S.C. Ematologia - Azienda Ospedali Riuniti Papardo-Piemonte, Messina, Italy
  - Unitа Linfomi - Dipartimento Oncoematologia, Istituto Scientifico San Raffaele, Milan, Italy
  - S.C. Ematologia - ASST Grande Ospedale Metropolitano Niguarda, Milan, Italy
  - Ematologia - A.O.U. Policlinico Giaccone, Palermo, Italy
  - Divisione di Ematologia - A.O. Ospedali Riuniti Villa Sofia-Cervello, Palermo, Italy
  - U.O. Ematologia - Ospedale Guglielmo da Saliceto, Piacenza, Italy
  - Ematologia - Azienda Unitа Sanitaria Locale-IRCCS - Arcispedale Santa Maria Nuova, Reggio Emilia, Italy
  - U.O. di Ematologia - Ospedale degli Infermi di Rimini, Rimini, Italy
  - Ematologia,Trapianto cellule staminali, Medicina Trasfusionale e Terapia cellulare -Policlinico Universitario Campus Bio-Medico, Roma, Italy
  - U.O.C. Ematologia - A.O.U. Senese, Siena, Italy
  - U.O.C. Ematologia - Ospedale di Circolo, Varese, Italy
  - Ospedale San Bassiano - AULSS7 Pedemontana - UOC Oncoematologia, Bassano del Grappa, Vicenza
  - Divisione di Oncologia e dei Tumori immuno-correlati - IRCCS Centro di Riferimento Oncologico di Aviano, Aviano